CLINICAL TRIAL: NCT05911594
Title: Efficacy and Safety of Intradetrusor BOTOX Injection Combined With Percutaneous Tibial Nerve Stimulation for Managing Children With Overactive Bladder Not Responding to Monotherapy
Brief Title: IDB Injection Combined With PTNS for Managing Children With OAB Not Responding to Monotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tamer Abd El-Wahab Diab, Lecturer of Urology, Faculty of Medicine, Benha University, Benha, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rc 14-2-2022
Record Dates: First submitted 2023-05-14; First posted 2023-06-22 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: BOTOX; Percutaneous Tibial Nerve Stimulation
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Solifenacin group (Experimental): Patients in this group will receive medical treatment (Solifenacin 5 mg once or twice daily) without any second line of treatment
  Interventions: Drug: Solifenacin group
- Percutaneous tibial nerve stimulation group (Experimental): Patients in this group will receive Percutaneous tibial nerve stimulation after failure of medical therapy
  Interventions: Procedure: Percutaneous tibial nerve stimulation group
- Intradetrusor BOTOX group (Experimental): Patients in this group will receive Intradetrusor BOTOX after the failure of medical therapy
  Interventions: Drug: Intradetrusor BOTOX group
- Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation group (Experimental): Patients in this group will receive Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation after the failure of medical therapy
  Interventions: Combination Product: Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation group

INTERVENTIONS:
Drug: Solifenacin group — Patients in this group will receive medical treatment (Solifenacin 5 mg once or twice daily) without any second line of treatment
  Arms: Solifenacin group
Procedure: Percutaneous tibial nerve stimulation group — Patients in this group will receive Percutaneous tibial nerve stimulation after failure of medical therapy
  Arms: Percutaneous tibial nerve stimulation group
Drug: Intradetrusor BOTOX group — Patients in this group will receive Intradetrusor BOTOX after failure of medical
  Arms: Intradetrusor BOTOX group
Combination Product: Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation group — Patients in this group will receive Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation after failure of medical
  Arms: Intradetrusor BOTOX combined with Percutaneous tibial nerve stimulation group

SUMMARY:
This study aimed to evaluate the outcome of simultaneous intradetrusor BOTOX (IDB) injection and Percutaneous tibial nerve stimulation (PTNS) for management of children with recurrent wetness since at least 6 months.

DETAILED DESCRIPTION:
Overactive bladder is a syndrome characterized by symptoms of urgency, with or without urgency incontinence, usually with increased daytime frequency and nocturia. The Neurogenic or myogenic bladder dysfunction can lead to the symptoms that characterize Overactive bladder. Normal bladder contraction occurs when the muscarinic receptors in the detrusor muscle are stimulated with acetylcholine. Although the pathogenesis of Overactive bladder is not fully explained; sensitization of afferent nerves, deactivation of inhibitory mechanisms, and the emergence of contractions similar to primitive voiding reflexes are shown as pathogenetic mechanisms. Another hypothesis is that the number of intercellular connections among detrusor myocytes increase, and these cells are spontaneously stimulated.

In addition to the fact that the etiopathogenesis cannot be explained clearly and due to the intense relationship with the autonomic nervous system, undesirable systemic side effects are common in treatments applied.

ELIGIBILITY:
Inclusion Criteria:

* Children with non-neurogenic overactive bladder defined after exclusion of neurogenic causes not responding to medical treatment for 6 months, and
* aged of 7-16 years
* presenting with recurrent night-time with occasional day-time wetness for overactive bladder.

Exclusion Criteria:

* recurrent OAB manifestations within less than 6 months after the previous monotherapy
* obstructive urinary tract diseases
* a history of pelvic surgery
* anatomical abnormalities
* neurogenic bladder
* syndromes that affect the bladder functions
* either current infection that was evidenced by urinalysis and culture or within the last two months
* systemic diseases inducing liability for wetness

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Overactive bladder symptom score | Baseline, 3, 6, 9 and 12 months after the intervention
  the Overactive bladder symptom score (OABSS) questionnaire will be calculated which consists of four items; namely, daytime frequency (score: 0-2), night-time frequency (score: 0-3), urgency (score: 0-5), and urgency incontinence (score: 0-5). The results scores were summed and a score of>8 suggesting an overactive bladder

SECONDARY OUTCOMES:
Patient Perception of Bladder Condition (PPBC) scale | Baseline, 3, 6, 9 and 12 months after the intervention
  The Patient Perception of Bladder Condition (PPBC) scale will be calculated which includes 6-point describing patient's comment of his/her bladder problems and ranging from 1: Not at all, 2: Some very minor, 3: Some minor, 4: some moderate, 5: severe, 6: many severe problems.
Patients' satisfaction | Up to the 12-month follow-up period
  The Patients' satisfaction will be assessed by the Likert scale (self-report scale where 0 = strong dissatisfaction, 1 = dissatisfaction, 2 = neutral, 3 = satisfaction, and 4 = strong satisfaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Urology departments Benha University Hospitals, Banhā, Qalyubiyya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The study will be available under a reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: One year after the end of the study